CLINICAL TRIAL: NCT01572519
Title: An Open-label, Multicenter, Phase 1/2 Study of JNJ-40346527, an FMS Inhibitor, in Subjects With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: A Study of JNJ-40346527 in Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100813; 40346527HKL1001 (Other: Janssen Research & Development, LLC); 2011-005795-42 (EudraCT Number)
Record Dates: First submitted 2012-02-16; First posted 2012-04-06 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Relapsed or Refractory Hodgkin Lymphoma
Keywords: Relapsed Hodgkin lymphoma; Refractory Hodgkin lymphoma; JNJ-40346527; Dose-escalation; Pharmacokinetics
MeSH Terms: conditions — Recurrence; Hodgkin Disease | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-40346527 (Experimental)
  Interventions: Drug: Phase 1, Cohort 1; Drug: Phase 1, Cohort 2; Drug: Phase 1, Cohort 3; Drug: Phase 1, Cohort 4; Drug: Phase 2

INTERVENTIONS:
Drug: Phase 1, Cohort 1 — Type=exact number, unit=mg, number=150, form=capsule, route=oral use. Capsule is taken once daily.
Drug: Phase 1, Cohort 2 — Type=exact number, unit=mg, number=300, form=capsule, route=oral use. Capsule is taken once daily.
Drug: Phase 1, Cohort 3 — Type=exact number, unit=mg, number=450, form=capsule, route=oral use. Capsule is taken once daily.
Drug: Phase 1, Cohort 4 — Type=exact number, unit=mg, number=600, form=capsule, route=oral use. Capsule is taken once daily.
Drug: Phase 2 — JNJ-40346527 at the recommended dose determined in Phase 1

SUMMARY:
The purpose of this study is to determine the safety, pharmacokinetics, and preliminary efficacy information of JNJ-40346527 in patients with relapsed or refractory Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is an open-label (individuals will know the identity of study treatments), dose-escalation study to evaluate the clinical efficacy, safety, and pharmacokinetics (PK; study of what the body does to a drug) of JNJ-40346527. Up to 38 subjects could be enrolled in the Phase 1 portion of the study and up to 30 subjects could be enrolled in the Phase 2 portion of the study (although planned, the study did not move forward to the Phase 2 portion). During the Phase 1 portion of the study, dose escalation of JNJ-40346527 will start at 150 mg (Cohort 1) once daily up to the maximum tolerated dose (MTD) or the highest planned dose (600 mg once daily); twice daily dosing may also be performed if deemed necessary. A Study Evaluation Team (SET) will review all available data after 1 cycle (21 days) of treatment for each cohort before any additional dose escalation occurs and will also determine the recommended Phase 2 dose for the expansion cohort. This study will consist of 3 periods: a screening period (from signing of informed consent until immediately before dosing), an open-label treatment period (from the first dose of study drug until the end-of-treatment visit), and a follow-up period (after the end-of-treatment visit). All patients will participate in the screening and treatment period. Patients will be administered JNJ-40346527 continuously until disease progression, or unacceptable toxicity (based on investigator assessment). The National Cancer Institute-Common Terminology Criteria for Adverse Events will be used to grade toxicity throughout the study. Disease response will be assessed according to the Revised Response Criteria for Malignant Lymphoma. Treatment will continue until disease progression or unacceptable toxicity (based on investigator assessment) occurs. Only patients who discontinue study drug before disease progression or discontinue due to treatment-related Grade 3 or higher toxicity will continue in the follow-up period. Serial PK samples will be collected in Cycle 1 as detailed in the protocol. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

- Patients with histopathologically confirmed initial diagnosis of Hodgkin lymphoma and who have disease that has relapsed or is refractory that is progressing or active and requires treatment after at least 1 appropriate therapy

Exclusion Criteria:

* Known brain metastases or leptomeningeal disease
* Other malignancy within past 5 years
* Has any condition that, in the opinion of the investigator, would make study participation not be in the best interest (eg, compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments
* QTc prolongation at screening or other factors that increase the risk of QT prolongation such as diagnosis or family history of long-QT syndrome, diagnosed or suspected congenital long QT syndrome, or concomitant use of medication that can prolong the QT interval
* Taking CYP3A4 substrate drugs with a narrow therapeutic index (eg, alfentanil, astemizole, sirolimus, tacrolimus, terfenadine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2013-08-13 (Actual); Study Completion 2013-08-13 (Actual)

PRIMARY OUTCOMES:
Phase 1 maximum tolerated dose (MTD) for JNJ-40346527 | After completion of Cycle 1 (21 days of dosing) in the last subject in Phase 1
Phase 2 overall response rate | Up to 6 months after the last subject is enrolled

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 6 months after the last subject is enrolled
Progression-free survival (PFS) | Up to 6 months after the last subject is enrolled
The number of participants affected by an adverse event | Up to 30 days after the last dose of study medication
Maximum observed plasma concentration of JNJ-40346527 | Up to treatment cycle Day 21
Trough plasma concentration of JNJ-40346527 | Up to treatment cycle Day 21
Minimum observed plasma concentration of JNJ-40346527 | Up to treatment cycle Day 21
Time of maximum observed plasma concentration of JNJ-40346527 | Up to treatment cycle Day 21
Area under the plasma concentration-time curve of JNJ-40346527 | Up to treatment cycle Day 21
Total drug clearance of JNJ-40346527 | Up to treatment cycle Day 21
Accumulation index of JNJ-40346527 | Up to treatment cycle Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- France (2):
  - Lille
  - Villejuif
- Germany (2):
  - Cologne
  - Würzburg

REFERENCES:
- See also: Link to results on EudraCT registry — https://www.clinicaltrialsregister.eu/ctr-search/trial/2011-005795-42/results